CLINICAL TRIAL: NCT05083234
Title: Maintaining Skin Integrity in Neonates With Sunflower Seed Oil and Liquid Vaseline: A Prospective Randomized Controlled Study
Brief Title: Maintaining Skin Integrity in Neonates With Sunflower Seed Oil and Liquid Vaseline
Acronym: Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Behice Ekici, Assistant Professor, PhD, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-10-01
Record Dates: First submitted 2021-10-04; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Neonatal Skin Conditions; Nursing Caries
Keywords: neonate; neonatal skin care; neonatal skin condition score; sunflower seed oil; liquid vaseline

STUDY DESIGN:
Intervention Model Description: Parallel Assigment,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sunflower Seed Oil Group (SSO) (Experimental): The skin of newborns in the sunflower seed oil group was moisturized with SSO
  Interventions: Other: Moisturizing with SSO
- Liquid Vaseline Group (LV) (Experimental): The skin of newborns in the liquid vaseline group was moisturized with LV.
  Interventions: Other: Moisturizing with LV
- Control Group (Experimental): The skin of newborns in the control group was not moisturized.
  Interventions: Other: The control group was not moisturized.

INTERVENTIONS:
Other: Moisturizing with SSO — Vital signs of newborns in the sunflower seed oil group were measured. The skin of newborns in the sunflower seed oil group was wiped without rubbing. The skin of newborns in the sunflower seed oil group was evaluated with the NSCS scale.
  Arms: Sunflower Seed Oil Group (SSO)
Other: Moisturizing with LV — Vital signs of newborns in the liquid vaseline group were measured. The skin of newborns in the liquid vaseline group was wiped without rubbing. The skin of newborns in the liquid vaseline group was evaluated with the NSCS scale.
  Arms: Liquid Vaseline Group (LV)
Other: The control group was not moisturized. — Vital signs of newborns in the control group were measured. The skin of newborns in the control group was wiped without rubbing. The skin of newborns in the control group was evaluated with the NSCS scale.
  Arms: Control Group

SUMMARY:
In this randomized controlled study, 90 preterm and term neonates in the NICU of a state hospital were equally divided into 3 groups. The skin integrity of the newborns in all three groups was assessed in terms of the Neonatal Skin Condition Score (NSCS), which was performed a total of 9 times at 48-hour intervals. The skin of the newborns in the first group was moisturized with SSO and with LV in the second group, once a day, a total of 17 times. Moisturizer was not applied to the skin of the third group of newborns (the control group).

DETAILED DESCRIPTION:
Because the barrier function of the skin of the newborn is still immature, disruption of skin integrity is a commonly observed problem. The purpose of the study was to test the applicability and effectiveness of sunflower seed oil (SSO) and Liquid Vaseline (LV) in maintaining skin integrity in term and preterm neonates in the Neonatal Intensive Care Unit (NICU). The sample size of the study has been determined by the power analysis (G*Power 3.1.9.2), The sample size was found to be a total of 66 neonates including minimum of 22 neonates for each group. It was estimated that case losses may occur and therefore, it was decided to conduct the study with a total of 90 neonates including 30 neonates in three groups. Assignment of neonates to research groups was done according to the order of hospitalization in the NICU. The first hospitalized neonates SSO, the second hospitalized LV, and the third hospitalized were included in the control group. The groups were repeated until they were complete. Weighing the neonate, taking vital signs, evaluating the skin condition, wiping the whole body, and stabilizing the general condition of the neonate before moisturizing the skin were taken into account. Neonates Information Form(NIF) and Neonatal Skin Condition Score (NSCS) were used for data collection. Parents of neonates were informed about the study. First day of hospitalization; Demographic data and medical history of the neonate in the study or control group were obtained from the patient file records. The neonate was weighed, vital signs were taken, and the data were recorded in the NIF.

The body of all neonates in the research or control group was wiped on the 1st day of hospitalization. In the following days, it was repeated 2 times a week (Monday and Friday) in the same way.The skin condition of the neonate in the research or control group was evaluated with the NSCS scale. The first skin evaluation was performed on the 1st day of hospitalization (1st NSCS). Skin condition was re-evaluated at 48 hour intervals in the following days. Skin condition of the neonate in the control or research group was evaluated a total of 9 times with 48-hour intervals. After the initial skin condition assessment, the neonate's skin is moistened with SSO or LV, depending on the group. It was rehydrated once a day (24 hours apart) in the following days.

ELIGIBILITY:
Inclusion Criteria:

* Parents giving verbal and written consent,
* Hospitalized in the NICU within the first 24 hours after birth,
* With a birth weight of more than 1500 g,
* No life-threatening health problems and skin diseases.

Exclusion Criteria:

* Gestational age less than 32 weeks,
* Parents who do not give verbal and written permission,
* Hospitalized in the NICU after the first 24 hours after birth,
* With a birth weight of less than 1500 g,
* Having life-threatening health problems and skin diseases.

Min Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Skin condition score of newborns | Change from skin condition score of newborns at 16 days
  The NSCS was developed for clinical nurses to use to evaluate infant skin condition. The scale evaluates skin dryness, erythema, and eruption. The best and worst possible scores are 3 and 9, respectively. The scale does not have a cutoff value. High scores indicate poor skin condition, and low scores indicate normal skin condition

CONTACTS AND LOCATIONS:
Overall Officials: Behice Ekici, PhD, Study Director — Maltepe University School of Nursing
Locations (1):
- Kanuni Sultan Süleyman Research and Training Hospital NICU, Istanbul, Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karakoc IB, Ekici B. Maintaining Skin Integrity in Neonates with Sunflower Seed Oil and Liquid Vaseline: A Prospective Randomized Controlled Study. Adv Skin Wound Care. 2022 Dec 1;35(12):1-8. doi: 10.1097/01.ASW.0000891080.13305.75. PMID 36409190